CLINICAL TRIAL: NCT06986421
Title: Perception of Post-stroke Patients, Physical and Rehabilitation Medicine Physicians, and Allied Health Professionals Regarding Advanced Rehabilitation Technology
Brief Title: Perception of Advanced Rehabilitation Technologies Among Post-Stroke Patients and Rehabilitation Staff
Acronym: P-TECH-AVC
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0378; 2025-A01110-49 (Other: ID-RCB)
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Post Stroke
Keywords: Rehabilitation; Stroke; Advanced Technology; Perception; Questionnaire
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Post-stroke patients: This group includes patients with a confirmed diagnosis of stroke, hospitalized or followed at HCL - Renée Sabran Hospital (Kermes 2 department), regardless of whether they have previously used advanced rehabilitation technologies.
  Interventions: Other: completion of a structured questionnaire
- Physicians in Physical and Rehabilitation Medicine: This group consists of physicians specialized in Physical and Rehabilitation Medicine, actively involved in the treatment and rehabilitation of post-stroke patients. Recruited from HCL - Renée Sabran Hospital and affiliated professional networks
  Interventions: Other: completion of a structured questionnaire
- Allied health professionals: This group includes allied health professionals involved in stroke rehabilitation, such as physiotherapists, occupational therapists, psychologists, speech therapists, neuropsychologists, and psychomotor therapists. All participants are affiliated with the HCL - Renée Sabran Hospital or collaborating institutions
  Interventions: Other: completion of a structured questionnaire

INTERVENTIONS:
Other: completion of a structured questionnaire — completion of a structured questionnaire

SUMMARY:
This observational study aims to assess the perception of advanced rehabilitation technologies among three key groups involved in stroke recovery: post-stroke patients, physicians specialized in Physical and Rehabilitation Medicine, and allied health professionals. The study is conducted at HCL - Renée Sabran Hospital , specifically within the Kermes 2 department. Participants are selected using a non-probability sampling method, based on predefined inclusion and exclusion criteria. Data will be collected using a structured, author-developed questionnaire designed to evaluate attitudes, perceived usefulness, ease of use, and intention to adopt technologies such as exoskeletons, social robots, wearable interactive devices, and biofeedback systems. The questionnaire is applied at a single time point after obtaining informed consent. This research responds to the growing integration of technology in neurorehabilitation and seeks to identify potential barriers or facilitators to its adoption in clinical practice.

The hypothesis is that there is a significant difference in perception and acceptance of advanced rehabilitation technologies between the three groups, influenced by their respective roles, experience, and level of exposure to such technologies.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Patients diagnosed with stroke, whether or not they have benefited from advanced rehabilitation technologies.
* Physicians: Physicians specialized in Physical and Rehabilitation Medicine who manage patients with stroke.
* Allied health professionals: Physiotherapists, psychologists, occupational therapists, speech therapists, neuropsychologists, and psychomotor therapists involved in the rehabilitation of post-stroke patients.

Exclusion Criteria:

* Refusal to participate in the study.
* Patients who do not wish to benefit from advanced rehabilitation technology.
* Healthcare professionals with no experience using advanced rehabilitation technologies.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from HCL - Renée Sabran Hospital, located in the PACA region (Provence-Alpes-Côte d'Azur), specifically from the Kermes 2 department, as well as through professional medical networks. The study population includes three main groups: (1) patients with a confirmed diagnosis of stroke, whether or not they have been exposed to advanced rehabilitation technologies; (2) physicians specialized in Physical and Rehabilitation Medicine involved in stroke management; and (3) allied health professionals (e.g., physiotherapists, psychologists, occupational therapists, speech therapists, neuropsychologists, psychomotor therapists) actively working in post-stroke rehabilitation settings. Recruitment will focus on individuals affiliated with institutions offering neurological rehabilitation services.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-07-08 (Estimated); Study Completion 2026-07-08 (Estimated)

PRIMARY OUTCOMES:
Perceptions of post-stroke patients, physical medicine and rehabilitation physicians and auxiliary medical staff on Advanced Rehabilitation Technologies. | Day 1
  The primary outcome measure evaluates the perception of advanced rehabilitation technologies among key stakeholders involved in post-stroke recovery. This perception is assessed using a structured questionnaire specifically developed by the authors, designed to capture attitudes, perceived usefulness, ease of use, and intention to adopt technologies such as exoskeletons, social robots, wearable interactive devices, and biofeedback systems. The instrument is applied to three target groups: post-stroke patients, physicians specializing in physical and rehabilitation medicine, and allied health professionals. This measure provides critical insights into the acceptability and potential integration of advanced technologies in neurorehabilitation practice.

CONTACTS AND LOCATIONS:
Overall Officials: David PLANTIER, DR, Principal Investigator — HCL
Locations (1):
- HCL - Renée Sabran Hospital, Hyères, France

IPD SHARING:
Plan to Share IPD: No